CLINICAL TRIAL: NCT05242575
Title: The Influence of Immersive Virtual Field Trips on Academic Vocabulary for Early Elementary Students With Developmental Language Disorder
Brief Title: The Influence of Immersive Virtual Field Trips on Academic Vocabulary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Salus University
Record Dates: First submitted 2022-01-23; First posted 2022-02-16 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2022-02

CONDITIONS: Developmental Language Disorder; Language Disorders in Children
Keywords: Developmental Language Disorder (DLD); Specific Language Impairment (SLI); Vocabulary
MeSH Terms: conditions — Language Development Disorders; Specific Language Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Book condition (No Intervention): Participants in the control condition will be receive a pre-recorded audio-visual book presentation. The purpose of pre-reading is to provide consistency in the examiner's affect and presentation, thereby controlling for potential examiner effects on study outcomes. Participants in the control group will receive three interventions each lasting 15-minutes. The number of sessions and intervention time is equal for both the control and experimental groups. The information provided in the control book and experimental iVFT parallel one another.
- Immersive virtual field trip (iVFT) (Experimental): The study intervention is a multisensory immersive virtual reality trip to the moon. Participants will use 3D cardboard goggles and a smart phone. No additional interventions will occur. Participants in the iVFT experimental group will receive three interventions each lasting 15-minutes. The number of sessions and intervention time is equal for both the control and experimental groups. Participants will explore the moon through a virtual reality scene by moving their body and head, which creates a 360º view. When hovering over items, participants are presented with several key elements related to word learning (e.g., written and spoken words/narrative). Multiple items are given extra emphasis through hotspots that provide audiovisual content in the form of brief videos and spoken scripts. The information provided in the iVFT and control book parallel one another.
  Interventions: Behavioral: The information provided in the iVFT and control book parallel one another.

INTERVENTIONS:
Behavioral: The information provided in the iVFT and control book parallel one another. — An immersive virtual fled trip (iVFT) is a form of virtual reality (VR). The term immersive refers to an experience where the senses become heightened through multisensory input (e.g., visual, auditory, proprioceptive). When adding peripherals such as a head-mounted device (HMD) (e.g., goggles with 3D-lenses), a mobile phone becomes a pseudo-theater providing a 360-degree view that mimics the real world. For example, one can experience a simulated rollercoaster or visit the moon that may otherwise be inaccessible in day-to-day life. Also, a VFT provides for context and aids in background knowledge that is a crucial aspect of learning.
  Participants will receive three interventions sessions each last 15-minutes.
  Other Names: Virtual Reality (VR)
  Arms: Immersive virtual field trip (iVFT)

SUMMARY:
The purpose of this study is to investigate an immersive virtual field trip (iVFT) on topic specific academic vocabulary for students with developmental language disorder (DLD). DLD is the most common childhood learning disorder with a prevalence of 7.4%(1) and occurs in the absence of a known biomedical condition (e.g., hearing loss, autism, stroke, intellectual disability). DLD affects a person's academic and social function due to difficulty with using and understanding language.(2,3) Approximately half of students with DLD have a deficit in vocabulary that persists through highschool.(4) Once children fall behind in their language and vocabulary development, it is very difficult to catch up generally resulting in a wider gap as they progress through their school years. This deficit can have cascading social, mental health, occupational and financial consequences.(5) There is preliminary evidence that a virtual reality experience such as an immersive virtual field trip (iVFT) was beneficial for facilitating vocabulary and comprehension in general education(6-8) and within targeted populations of students including second language learners(9) and those with learning differences (e.g., autism,(10) attention deficit hyperactivity,(11,12) and dyslexia(13). The term "immersive" refers to a state of heightened sensation when viewing a simulated environment that is superimposed onto a screen with embedded multisensory input (e.g., visual, auditory, proprioceptive).(14) The viewer looks through 3D goggles to block out the present environment resulting in a feeling of presence. These simulated experiences or destinations (e.g., space) are a type of VR referred to as an immersive virtual field trip (iVFT).

To date, there is a lack of empirical evidence, explicitly targeting academic vocabulary growth for early grade school students with DLD. In addition, no study has reported on learning outcomes of students with DLD following a VR condition. Therefore, the primary study objective was to compare gains in academic vocabulary measures between a traditional book condition and an iVFT learning condition for young students with DLD.

DETAILED DESCRIPTION:
The purpose of this randomized control study is to investigate an immersive virtual field trip (iVFT) for learning academic vocabulary for students with developmental language disorder (DLD).

The primary objective is to compare gains in topic specific vocabulary measures between a traditional book condition and an iVFT learning condition. Also, this study will compare perceptions of the study experience between the control and experimental groups.

At study entry, 24 children between the ages of 6:0 to 8:12 years old with a developmental language disorder (DLD) will be randomized to equal groups of control book and experimental iVFT conditions.

If satisfy the inclusion and exclusion criteria, a three-phase pre-enrollment process will ensue. In the first phase, the Student Language Scale (SLS) and Shaywitz Dyslexia screeners will be administered to determine likelihood of presence of a language disorder and functional impact on academic and social growth. In the second phase, the CELF-5 diagnostic language assessment will determine the presence of a DLD if a standard score equal or less than 75 is obtained. In the third phase, the PPVT-5 vocabulary assessment will be administered to provide additional information about general receptive vocabulary knowledge. Lastly, four topic specific vocabulary measures will provide a measure of baseline topic vocabulary knowledge.

Consented and enrolled participants will be randomized into equal groups of control and experimental conditions. The control group will receive a pre-read book and the experimental group will be exposed to an immersive virtual field trip using 3D cardboard goggles and a smart phone. The content in the book and iVFT parallel one another. In both groups, audio and visual stimuli are presented. For all participants, a total of three 15-minute exposures will occur.

Following the condition, the four-topic specific vocabulary measures will be repeated to report on vocabulary growth. The measures include:

1. Divergent Naming (expressive): "Tell me the names of as many [topic] as you can think of, as quickly as possible, in one minute."
2. Word Naming (expressive confrontational naming): State name of target image presented in isolation.
3. Picture Identification (receptive): Identify target picture in field of ten.
4. Word meaning recognition: Match the word with the written meaning. Lastly, all participants will rate experience their experience using an Intrinsic Motivation Inventory (IMI) with a 5-point Smile Likert Scale.

The data analysis will include descriptive and inferential statistics to report within and between group gains in the four-topic specific vocabulary measures.

ELIGIBILITY:
Inclusion Criteria:

* Age 6.0- 8.12 years.
* English language proficiency determined by examiner screening.
* Spoken language is readily understandable by examiner.
* Child speaks at least five-word sentences per examiner screening.
* Child understands and can follow two-part directions per examiner screening.
* Subject can complete all study protocol assessments.
* Sees single image in binoculars and sees 3D images.
* Diagnosis of developmental language disorder (DLD) (determined by ≤-1SD on the Clinical Evaluation of Language Fundamentals (CELF-5) completed within the past 12 months or examiner evaluation with the CELF-5.
* Vocabulary deficit determined by scores equal to or less than 30% on two or more topic specific vocabulary measures.
* Access to home Wi-Fi with sufficient connectivity to run the iVFT
* VFT compatible smartphone to include operating systems iOS 8.0 (e.g., Apple iPhone 6 or later) or later or Android 4.1 (JellyBean) or later (e.g., Samsung Galaxy S5 or later).

(Note: If a participant would otherwise not be able to participate, a loaner device will be provided to the parent/guardian for study purposes.)

Exclusion Criteria:

* History of the following medical conditions

  * Seizures/epilepsy
  * Moderate to severe motion sickness, cybersickness
  * Vision impairment defined as any child who has 504 plan requiring accommodations for visual impairment
  * Hearing impairment that prevents a child from hearing audio on a mobile device, a history of a failed hearing screening that has not been resolved, or a hearing impairment that results in an educational impact and requires specially designed instruction under IDEA (34 CFR § 300.8)."
* Inability to use the smart phone application
* Classified by school district as LEP (limited English proficient).
* Children who are wards of the state or any other agency, institution, or entity will not be solicited for participation.
* Intellectual disability (based on IEP/504 status).

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Compare vocabulary gains between the book and iVFT conditions | 1 week: pretest, three 15-minute intervention sessions, posttest
  Change in target vocabulary words from pre to post intervention between the control book condition and the iVFT learning condition. Four-topic specific omnibus vocabulary measures include:
  1. Divergent Naming (expressive): "Tell me the names of as many [topic] as you can think of, as quickly as possible, in one minute." One point earned for each named word.
  2. Word Naming (expressive confrontational naming): State name of target image presented in isolation. One point earned for each correct response.
  3. Picture Identification (receptive): Identify target picture in field of ten. One point earned for each correct response.
  4. Word meaning recognition: Match the word with the written meaning. One point earned for each correct response.

SECONDARY OUTCOMES:
Vocabulary growth following an iVFT condition | 1 week: pretest target vocabulary, three 15-minute intervention sessions, posttest target vocabulary
  To determine if an iVFT is effective for improving topic-specific vocabulary four omnibus vocabulary measures will be conducted pre-treatment and re-administered post-treatment.
  omnibus vocabulary measures include:
  1. Divergent Naming (expressive): "Tell me the names of as many [topic] as you can think of, as quickly as possible, in one minute." One point earned for each named word.
  2. Word Naming (expressive confrontational naming): State name of target image presented in isolation. One point earned for each correct response.
  3. Picture Identification (receptive): Identify target picture in field of ten. One point earned for each correct response.
  4. Word meaning recognition: Match the word with the written meaning. One point earned for each correct response.
Compare group perceptions of the study experience. | 1 week: following three 15-minute intervention sessions
  Following post vocabulary testing, participants will rate their experience by responding to a 15 question Intrinsic Motivation Inventory (IMI) with a 5-point Smile Likert Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Scheiman, PhD, DO, Study Chair — Dean of Research; Amy Lustig, PhD,SLP,MPH, Study Chair — Salus Univeristy; Yvonne D'Uva Howard, PhD, MS SLP, Principal Investigator — Salus University
Locations (1):
- Salus University, Elkins Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared